CLINICAL TRIAL: NCT01882517
Title: The Cholesterol Lowering Efficacy of Plant Stanol Ester Yoghurt in a Turkish Population
Brief Title: Lipid-lowering Effect of Plant Stanol Yogurt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Raisio Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCL_2010_024
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Hypercholesterolemia; Hyperlipidemias; Dyslipidemias
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yogurt that contains plant stanol esters (Active Comparator): Dietary Supplement: Yogurt that contains plant stanol esters
  Interventions: Dietary Supplement: Yogurt that contains plant stanol esters
- Placebo yogurt (Placebo Comparator): Dietary Supplement: Placebo yogurt
  Interventions: Dietary Supplement: Placebo yogurt

INTERVENTIONS:
Dietary Supplement: Yogurt that contains plant stanol esters
  Arms: Yogurt that contains plant stanol esters
Dietary Supplement: Placebo yogurt
  Arms: Placebo yogurt

SUMMARY:
To determine the effect of investigational products on serum LDL cholesterol.

DETAILED DESCRIPTION:
Efficacy of plant stanols as esters on LDL-cholesterol reduction is well documented. LDL-cholesterol lowering efficacy of the ingredient administered in a yogurt is less well known.

Study was monitored by Foodfiles

ELIGIBILITY:
Inclusion Criteria:

* subjects must voluntarily sign the informed consent
* subjects must be male or female aged 20 to 70 years
* subjects must have a serum total cholesterol concentration of 5.2 - 7.5 mmol/l ( 205 - 290 mg/dl) at the screening visit (visit 1, -2 week)

Exclusion Criteria:

* subjects using lipid lowering medication
* subjects using ezetimibe
* subjects with bile acid sequestrant medication
* subjects with statin therapy
* subjects using other medication significantly influencing on lipid values
* subjects with diagnosis type 1 or type 2 diabetes
* severe obesity (BMI>35.0 kg/m2)
* serum fasting triglycerides > 4.0 mmol/l
* subjects with any hepatic or renal disorder according to medical history
* subjects who have history of myocardial infarction or unstable angina pectoris within six months prior to screening
* subjects who have history of coronary artery bypass graft or percutaneous transluminal coronary angioplasty within six months prior to screening
* subjects who have history of temporal ischemic attack or stroke within six months prior to screening
* subjects who have a history of cancer or other malignant disease within the past five years
* subjects with abnormal values of health screening variables measured at screening visit: serum gamma-glutamyltransferase> 2 x upper limit, serum alkaline phosphatase> 2 x upper limit or other abnormality in laboratory evaluations considered as clinically significant in the opinion of the study physician
* subjects who are consuming more than 15 portions of alcohol / week
* subjects who are pregnant or lactating
* subjects using Benecol, Becelpro.activ, Danacol or other plant sterol enriched products within 30 days before visit 2
* subjects with severe lactose intolerance, milk allergy or any other intolerance to the ingredients of test products
* celiac disease

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-03; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in serum LDL cholesterol | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)